CLINICAL TRIAL: NCT07397780
Title: RPMO2 Oximeter Accuracy During Sleep 1 Trial
Acronym: ROADS-1
Status: Recruiting | Type: Observational
Sponsor: ProSomnus Sleep Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: SP-008
Record Dates: First submitted 2026-01-26; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; oral appliance therapy; mandibular advancement; oximetry
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: RPMO2 OSA Device — Buccal mucosal oximeter embedded into the upper dental arch of an oral appliance used to treat obstructive sleep apnea.

SUMMARY:
The goal of this observational study is to validate the accuracy of the RPMO2 OSA Device's oxygen desaturation index in individuals with obstructive sleep apnea versus the gold standard, in-lab polysomnography.

Participants will receive an RPMO2 OSA Device and complete one night in a sleep lab using the device in addition to the standard montage used for polysomnography.

DETAILED DESCRIPTION:
Monitoring of physiologic variables indicative of the presence and status of chronic disease have proven to be of considerable value in the clinical management and improvement of therapeutic outcomes. For instance, positive airway pressure (PAP) devices used in the treatment of obstructive sleep apnea (OSA) and pulmonary diseases provide nightly monitoring of therapeutic pressures and pulmonary disturbances. Sleep-related declines in the oxyhemoglobin saturation of arterial blood (SaO2) are a common and important pathophysiological occurrence and are associated with cardiovascular incidences and decreased survival in patients with sleep apnea. As well, such nocturnal hypoxia displays substantial night-to-night variability in respiratory status during sleep. Thus, the need for a comfortable, accurate oximeter capable of multi-night monitoring seems undeniable. Nonetheless, standard pulse oximeters are not commonly used for multi-night monitoring of SaO2 as the currently available devices are cumbersome and disturb sleep. An important consideration is that nightly monitoring must be convenient and inexpensive, features not present in currently available oximeters. The accuracy of conventional oximeters can be compromised by factors such as movement, poor perfusion, impaired thermoregulation, and ambient light interference. Importantly, SpO2 readings have been shown to be overestimated in individuals with darker skin, potentially leading to increased incidence of occult hypoxemia.

ProSomnus Sleep Technologies (Pleasanton, CA, USA) has developed a novel buccal mucosal oximeter (RPMO2 OSA Device). The oximeter is encapsulated in an overlay of the maxillary dentition and uses the mucosa of the buccal vestibule behind the upper lip as the reflective tissue. This device is suitable for long-term nightly monitoring as it is comfortable and rechargeable. Additionally, the site of the oximeter sensor, the buccal mucosa, has the advantages of being highly vascular, relatively void of melanin, and protected from ambient light. The device has been validated in a controlled desaturation study per ISO 80601-2-61, in which arterial blood samples from healthy, awake volunteers were collected and analyzed using co-oximetry while volunteers were desaturated from ~97% to ~72% SaO2. The RPMO2 device met the accuracy requirements stipulated by the United Stated Food and Drug Administration for reflectance pulse oximeters, i.e., ARMS ± 3.5% for SpO2 and ARMS ± 3bpm for pulse rate.

The purpose of the present investigation is to validate the accuracy of the RPMO2 device in adults with OSA during sleep versus the gold standard, in-lab polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 years or older
* Diagnosed with obstructive sleep apnea (per American Academy of Sleep Medicine's definition)
* Adequate dentition for oral appliance therapy
* Ability to refrain from the use of OSA therapy other than the study device for the week prior to the in-lab sleep study

Exclusion Criteria:

* Non-respiratory sleep disorders or environmental or personal factors that preclude the accuracy, acquisition, or interpretation of in-lab polysomnography
* Pregnancy
* In the opinion of the principal investigator, unsuitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with obstructive sleep apnea
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Agreement between 4% oxygen desaturation index between study device and polysomnography | 1 week
  The primary study endpoint is the paired difference in 4% ODI between the study device and polysomnography (PSG). A paired design will be used to test agreement of 4% ODI as measured using the study device and manually scored PSG simultaneously. The Bland-Altman 95% limits of agreement (LoA) and their 95% confidence intervals (CI) for the LoA will be calculated. The maximum absolute value of the CIs will be compared to the maximum allowable difference. Agreement will be concluded if the maximum absolute value of the CIs is < 19.

CONTACTS AND LOCATIONS:
Locations (1):
- Star Sleep and Wellness, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No